CLINICAL TRIAL: NCT02795234
Title: Empirical Comperative Study Of Variation Blood Level Antibody Vitamin D at Different Groups Of Patients Compared Healthy Peoples And The Correlation Between Vitamin D Level
Brief Title: Empirical Comperative Study Of Variation Blood Level Antibody Vitamin D at Different Groups Of Patients Compared Healthy Peoples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, Head of Internal Medicine, Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Vitamin D 25 - 2016
Record Dates: First submitted 2016-06-05; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants with Vitamin D deficiency (Other): Blood sample, venous blood, about 10 ml will be drawn from participants and tested for the presence of Vitamin D antibodies
  Interventions: Other: Blood samples
- Participants with sufficient Vitamin D Level (Other): Blood sample, venous blood, about 10 ml will be drawn from participants and tested for the presence of Vitamin D antibodies
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
The aim of this study is to detect antibodies to vitamin D in the serum at Different Groups of patients and healthy volunteer. A second goal is to find the relation between Vitamin D Antibody and Vitamin D level.

DETAILED DESCRIPTION:
Vitamin D and its metabolites have a significant role in the calcium homeostasis and bone metabolism. Vitamin D deficiency as measured by serum 25(OH)D below 20 ng/mL (50 nmol/L) may contribute to the development of osteoporosis and Osteomalacia.

Several studies have clearly demonstrated that low 25(OH)D levels are associated with more comorbidities, higher estimated cardiovascular risk and autoimmune diseases.

Exposure to the ultraviolet (UV) rays in sunlight is the major source of vitamin D. other sources are dairy products enriched with vitamin D.

Vitamin D deficiency can result from inadequate exposure to sunlight, malabsorption including inflammatory bowel disease, celiac disease and patients undergone resection of the small intestine and inadequate intake of dairy products enriched with vitamin D.

Another possible explanation for vitamin D deficiency is the presence of neutralizing autoantibodies to vitamin D.

The aim of this study is to detect antibodies to vitamin D in the serum at Different Groups of patients and healthy volunteer

At least 64 Blood samples of Patients and healthy volunteer will be tested for the presence of auto-antibodies using an ELISA reader.

The result will compare antibody-positive and antibody-negative individuals with respect of serum 25(OH)D level and other variables and to find the relation between Vitamin D Antibody and Vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated in Meir Medical Center
2. Data on serum vitamin D values
3. 18 years old
4. Both sexes
5. Patient hereby declare that he\she agree to participate the clinical trial

Exclusion Criteria:

1. Patient refuses to sign Informed Consent.
2. Patients without vitamin D values

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Presence of Anti Vitamin D Antibodies in Blood Sample | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: reut ohanah, Principal Investigator — Meir Medical Center